CLINICAL TRIAL: NCT06825884
Title: Use of Extracellular Vesicles (EV) for Diabetic Foot Ulcers
Acronym: EVDFUUJCTC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Abdalla Awidi Abbadi, MD (Unknown)
Responsible Party: Principal Investigator, Hanan Jafar, Principal Investigator, University of Jordan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVDFUUJCTC; University of Jordan (Other: Cell Therapy Center)
Record Dates: First submitted 2025-01-23; First posted 2025-02-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Extracellular micro vesicles (EV) as direct perilesional injection into the diabetic chronic foot ulcers (DFU) which have not healed after using standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracellular vesicles (EV) (Experimental): * Patients will receive 5 ml perilesional injections as treatment weekly interval.
  * Post injection dressing will be with exofiber and bandaging.
  * Off-loading will apply when required.
  * Quantitative ulcer healing will be calculated according the surface area of the remaining ulcer at week 10 and12.
  * Standard of care will be given throughout the whole study period from week 1 through week 12.
  Interventions: Biological: Extracellular micro vesicles (EV)

INTERVENTIONS:
Biological: Extracellular micro vesicles (EV) — Extracellular micro vesicles (EV) as direct perilesional injection into the diabetic chronic foot ulcers (DFU) which have not healed after using standard of care.

SUMMARY:
Diabetes Mellitus is a common chronic medical condition that requires complex care strategies. Treatment includes methods to reduce glycemic burden and maintain glycemic control in the patient to prevent symptoms of hyperglycemia and reduce microvascular complications. In the case of patients with diabetes mellitus, wound healing, skin re- epithelization and skin integrity restoration are compromised, leading to chronic cutaneous ulcers such as diabetic foot ulcers. As much as 15% of all diabetic patients manifest diabetic foot ulcers. Moreover, 84% of all diabetes related lower leg amputations are anticipated to the result of diabetic foot ulcers. Compromised chronic cutaneous ulcer healing may result from cytokines, growth factor deficits, and insufficient angiogenesis process.

DETAILED DESCRIPTION:
Diabetes Mellitus is a common chronic medical condition that requires complex care strategies. Treatment includes methods to reduce glycemic burden and maintain glycemic control in the patient to prevent symptoms of hyperglycemia and reduce microvascular complications. In the case of patients with diabetes mellitus, wound healing, skin re- epithelization and skin integrity restoration are compromised, leading to chronic cutaneous ulcers such as diabetic foot ulcers. As much as 15% of all diabetic patients manifest diabetic foot ulcers. Moreover, 84% of all diabetes-related lower leg amputations are anticipated to be the result of diabetic foot ulcers. Compromised chronic cutaneous ulcer healing may be ascribed to cytokines, growth factor deficits, and insufficient angiogenesis process.

Wound healing is a process that begins as a reaction to skin injury, re-epithelization is a crucial phase of the wound healing, and it is impelled by keratinocytes migration and proliferation. Cell migration and proliferation are initiated and regulated by growth factors and cytokines that are released from the wounded epithelium. Restoration of skin integrity in the case of chronic cutaneous ulcers in patients with diabetes mellitus is compromised. Autologous human platelet granules, such as human platelet lysate (hPL) and extracellular micro vesicles (EV), represent a promising source of bioactive substances and have shown to be effective both in vitro and in vivo in wound healing studies. Prior studies supported the use of platelet rich plasma and extracellular micro vesicles in healing chronic lower extremity wounds and the treatment of diabetic foot ulcers.

The investigators are proposing this work for the use of bioactive substance:

Extracellular micro vesicles (EV) as direct perilesional injection into the diabetic chronic foot ulcers (DFU) which have not healed after using standard of care. This is a clinical study in chronic DFU stage A2 and A3 as per the university of Texas DFU classification (Appendix I), corresponding to Wegner classification III; IV.

ELIGIBILITY:
Inclusion Criteria:

Persons with type 2 diabetes between the ages of 30 and 75 with an ulcer of at least 6 weeks' duration. 2. Hemoglobin A1C< 11. 3. Index foot ulcer located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces); and wound area (length x width) measurement between 1 cm 2 and 60 cm 4. Wounds located under a Charcot deformity should be free of acute changes and must have undergone appropriate structural consolidation. 5. The index ulcer should be clinically non-infected and full-thickness without exposure of bone. 6. The protocol requires that post debridement; the ulcer would be free of necrotic debris, foreign bodies or sinus tracts. 7. Non- invasive vascular testing ankle brachial pressure index (ABPI) < 0.80. 8. Physical examination (including a Semmes-Weinstein monofilament test for neuropathy using the 5.07/10 g monofilament to test the plantar aspects of the great toe, third, and fifth metatarsal heads. 9. Negative for infectious panel (HIV, HBV, HCV, and VDRL). 10. Approved signed informed consent. 11. Coding and Randomization.

Exclusion Criteria:

1. Patient currently enrolled in another investigational device or drug trial or previously enrolled (within last 30 days) in investigative research of a device or pharmaceutical agent.
2. Ulcer decreased (up to) 25% in area during 7-day screening period.
3. Ulcer is due to non-diabetic etiology.
4. Patient's blood vessels are non-compressible for ABI testing.
5. Evidence of gangrene in ulcer or on any part of the foot.
6. Patient has radiographic evidence consistent with diagnosis of acute Charcot foot.
7. Patient is currently receiving or has received radiation or chemotherapy within 3 months of treatment.
8. Patient has received growth factor therapy within 7 days of treatment.
9. Screening hemoglobin <10.0 mg/dL.
10. Screening platelet count < 100 x 10 9 /L.
11. Patient is undergoing renal dialysis, has known immune insufficiency, known abnormal platelet activation disorders, eating/ nutritional, hematologic, collagen vascular disease, rheumatic disease, or bleeding disorders.
12. History of peripheral vascular repair within the 30 days.
13. Patient has known or suspected osteomyelitis.
14. Surgical correction (other than debridement) required for ulcer to heal.
15. Index ulcer has exposed bone.
16. Patient is known to have a psychological, developmental, physical, emotional, or social disorder, or any other situation that may interfere with compliance with study requirements and/or healing of the ulcer.
17. History of alcohol or drug abuse within the last year prior to randomization.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
To determine the short-term speed and effectiveness of extracellular micro vesicles (EV) on the healing of diabetic foot ulceration. And to prove that extracellular micro vesicles (EV) will significantly shorten the required timeto heal DFU. | follow-up duration is 12 months
  After measuring the wound area surface
  * the investigators will consider that the wound is full-healed when its surface area is healed (100%)
  * the investigators will consider that the wound is partial-healed when its surface area is healed (50- 100%)
  * the investigators will consider that the wound is minimal-healed when its surface area is healed (25- 50%)
  * the investigators will consider that the wound is non-healed when its surface area is <25%

CONTACTS AND LOCATIONS:
Locations (1):
- Cell Therapy Center, Amman, Jordan